CLINICAL TRIAL: NCT04611932
Title: A Randomized, Open-label, Single Dose, 3-period Partial Replicated Crossover Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-333 Low Dose in Healthy Volunteers Under Fasting Conditions
Brief Title: Clinical Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-333 Low Dose in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A70_08BE1907
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reference-Reference-Test (Experimental)
  Interventions: Drug: CKD-330 Tab. and D090 Tab.; Drug: CKD-333 Tab.
- Reference-Test-Reference (Experimental)
  Interventions: Drug: CKD-330 Tab. and D090 Tab.; Drug: CKD-333 Tab.
- Test-Reference-Reference (Experimental)
  Interventions: Drug: CKD-330 Tab. and D090 Tab.; Drug: CKD-333 Tab.

INTERVENTIONS:
Drug: CKD-330 Tab. and D090 Tab. — 1T
  Other Names: Reference
Drug: CKD-333 Tab. — 1T
  Other Names: Test

SUMMARY:
This study is a randomized, open-label, single dose, 3-period partial replicated crossover study to evaluate the pharmacokinetic profiles and safety of CKD-333 low dose in healthy volunteers under fasting conditions.

DETAILED DESCRIPTION:
To healthy subjects of fifty-one (51), following treatments are administered dosing in each period and wash-out period is a minimum of 14 days.

Reference drug: 1) Cantabell Tab. 8/5mg 2) Lipitor Tab. 10mg / Test drug: CKD-333 8/5/10mg Tab.

Pharmacokinetic blood samples are collected up to 72hrs. The pharmacokinetic characteristics and safety are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults over the age of 19 years and under the age of 55 years at the time of screening
2. Individuals who had 17.5 kg/m2 ≤ Body Mass Index(BMI) < 30.5kg/m2 and men's total body weight ≥ 55 kg, women's total body weight ≥ 45 kg

   * BMI = Weight(kg)/ Height(m)2
3. Individuals without congenital/chronic diseases and without abnormal symptoms or diagnosis based on a medical examination within the last 3 years
4. Individuals who were deemed to be appropriate as study subjects following laboratory tests (hematology, blood chemistry, urinalysis, viral/bacterial, etc.) and vital signs, ECG etc. performed at screening
5. Individuals who signed an informed consent form approved by the IRB of Chonbuk National University Hospital and decided to participate in the study after being fully informed of the study prior to participation, including the objective, content and characteristics of the investigational product
6. Individuals who agreed proper contraception during the study and did consent to not donation of sperm 1 month after the last dose of study drug infusion
7. Individuals with the ability and willingness to participate the entire study period

Exclusion Criteria:

1. Individuals with a medical evidence or a history (excluding a dental history of periodontal surgery, impacted wisdom teeth removal, etc.) of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurologic or immune diseases.
2. Individuals with a medical history of gastrointestinal disease (e.g., gullet disease such as esophageal achalasia and esophagostenosis and Crohn's disease) or operations (excluding simple appendectomy, herniotomy or tooth extraction) that may affect drug absorption
3. Individuals with the following laboratory test results at screening:

   * ALT or AST > 2x the upper limit of the normal range
   * CK > 3x the upper limit of the normal range
4. History of regular alcohol consumption exceeding 210 g/week within the 6 months prior to screening (1 drink (250 mL) of beer (5%) = 10 g; 1 drink (50 mL) of hard liquor (20%) = 8 g; 1 drink (125 mL) of wine (12%) = 12 g)
5. Individuals who smoked more than 20 cigarettes per day within 6 months prior to screening
6. Individuals who had been administered investigational product(s) from other clinical study or bioequivalence study within the 6 months prior to the first dose of this study
7. Following vital signs results at screening

   - Sitting systolic blood pressure ≥ 140 mmHg or < 90 mmHg and/or sitting diastolic blood pressure ≥90 mmHg or <60 mmHg
8. Individuals with a medical history of significant alcohol or drug abuse within one year prior to the screening
9. Individuals who had taken any drug(s) known as a strong inducer(s) or inhibitor(s) of drug-metabolizing enzymes within 30 days prior to the first dose of investigational product(s)
10. Individuals who had taken prescription or nonprescription drugs within the 10 days prior to the first dose of investigational product(s)
11. Individuals who donated whole blood within the 2 months, or blood components within 1 month prior to the first dose of the investigational product(s)
12. Individuals with severe acute/chronic medical or psychiatric condition that may increase the risk associated with study participation or investigational product(s) administration, or may interfere with the interpretation of study results
13. Individuals with hypersensitivity to investigational products or the investigational products ingredients or dihydropyridine drugs
14. Patient with hyperkalemia
15. Patients with hepatopathy
16. Patients with hereditary angioedema, ACE inhibitors or angiotensin Ⅱ receptor antagonists who have a history of angioedema
17. Primary hyperaldosteronism
18. Patients with aortic valve stenosis, mitral (valve) stenosis, hypertrophic obstructive cardiomyopathy
19. Patients with ischemic heart disease, ischemic cardiovascular disease, cerebrovascular disease
20. Patients with Intravascular volume depletion
21. Patients with nephropathy (eGFR<60 ml/min/1.73 m2)
22. Patients with renal artery stenosis
23. Patients with muscle disease
24. Patients with Hypothyroidism
25. Women who are pregnant or may be pregnant
26. Patients with a history of muscle toxicity when using statins or fibrates
27. Patients who are taking glecaprevir/pibrentasvir
28. Patients with hereditary diseases of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption etc.
29. Individuals who were deemed to be inappropriate to participate in the study by the investigator

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2020-11-11 (Estimated); Primary Completion 2021-03-10 (Estimated); Study Completion 2021-04-27 (Estimated)

PRIMARY OUTCOMES:
AUCt of CKD-330, D090, CKD-333 | Pre-dose (0 hour), post-dose 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  Area under the CKD-330/D090/CKD-333 concentration in blood-time curve from zero to final
Cmax of CKD-330, D090, CKD-333 | Pre-dose (0 hour), post-dose 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  The maximum CKD-330/D090/CKD-333 concentration in blood sampling time t

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No